CLINICAL TRIAL: NCT02716311
Title: Phase II Study Evaluating the Combination of Cetuximab With Afatinib as First-line Treatment for Patients With EGFR Mutated Non Small Cell Lung Cancer
Brief Title: Combination of Cetuximab With Afatinib for Patient With EGFR Mutated Lung Cancer
Acronym: ACE-Lung
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Intergroupe Francophone de Cancerologie Thoracique (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IFCT-1503
Record Dates: First submitted 2015-11-30; First posted 2016-03-23 (Estimated); Last update posted 2022-08-11 (Actual); Status verified 2022-08

CONDITIONS: Non Small Cell Lung Cancer
Keywords: EGFR; Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms | interventions — Afatinib; Cetuximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Afatinib (Other): Afatinib 40 mg/d until progression
  Interventions: Drug: Afatinib
- Afatinib + cetuximab (Experimental): Afatinib 40 mg/d until progression + cetuximab 500 mg/m² every 2 weeks during 6 months (beginning at D15 at 250 mg/m²)
  Interventions: Drug: Afatinib; Drug: Cetuximab

INTERVENTIONS:
Drug: Afatinib
Drug: Cetuximab
  Arms: Afatinib + cetuximab

SUMMARY:
Until recently, the first line treatment of metastatic Non Small Cell Lung Cancer (NSCLC) was a platine-based chemotherapy. It has been changed by the discovery of EGFR (Epidermal Growth Factor Receptor) mutations and associated treatment with Tyrosine Kinase Inhibitor (TKI) of EGFR. The superiority of EGFR TKI over chemotherapy for EGFR mutated patients has been proved in several phase III trials with gefitinib, erlotinib or afatinib.

Nevertheless, all patients will progress after 9 to 12 months of treatment due to the appearance of a treatment resistance.

Afatinib is an irreversible EGFR TKI. It binds to its receptor permanently.Contrary to erlotinib and gefitinb which inhibits only EGFR, afatinib inhibits the kinase activity of all HER family (Human Epidermal growth factor Receptor). Nevertheless, there is no proof that afatinib delay the appearance of resistance.

Cetuximab is a monoclonal antibody which binds specifically with EGFR. The double inhibition of EGFR by afatinib and cetuximab has demonstrated its efficacy in pre-clinical models. The hypothesis of this study is that the combination between cetuximab and afatinib will permit to delay or decrease the appearance of resistances.

ELIGIBILITY:
Principal Inclusion Criteria:

* Stage III or IV NSCLC, non irradiable non operable
* Non squamous NSCLC histologically or cytologically confirmed
* No previous treatment of NSCLC
* EGFR mutation (exon 19 deletion, L858R mutation, G719X , L861Q or S768I mutations or exon 19 insertion)
* Presence of at least one lesion that can be measured
* PS 0 or 1

Principal Exclusion Criteria:

* Symptomatic brain metastasis or requiring immediate radiotherapy
* T790M mutation or exon 20 insertion
* Radiotherapy less than 2 weeks prior randomization including symptomatic radiotherapy
* Interstitial pneumopathy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 118 (Actual)
Dates: Start 2016-05 (Actual); Primary Completion 2019-02 (Actual); Study Completion 2021-04-07 (Actual)

PRIMARY OUTCOMES:
Time to Treatment Failure | 9 months

SECONDARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | 1 month
Response Rate | 9 months
Overall survival | 6 months
Overall survival | 9 months
Overall survival | 12 months
Progression-Free Survival | 6 months
Progression-Free Survival | 9 months
Progression-Free Survival | 12 months
Progression-Free Survival | 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Alexis CORTOT, MD, PhD, Principal Investigator — CHRU LILLE; Jacques CADRANEL, MD, PhD, Principal Investigator — AP-HP Hôpital Tenon, Paris
Locations (33):
- France (33):
  - Centre Hospitalier du Pays d'Aix, Aix-en-Provence
  - Clinique de L'Europe, Amiens
  - Angers - CHU, Angers
  - Annecy - CH, Annecy
  - Bordeaux - Institut Bergonié, Bordeaux
  - Bordeaux - Polyclinique Nord, Bordeaux
  - Boulogne - Ambroise Paré, Boulogne-Billancourt
  - Clermont-Ferrand - CHU, Clermont-Ferrand
  - CH, Colmar
  - CHRU Grenoble, Grenoble
  - Centre Hospitalier - Pneumologie, Le Mans
  - CHRU de Lille, Lille
  - Lille - Polyclinique de la Louvière, Lille
  - Lyon - Hôpital Privé Jean Mermoz, Lyon
  - Institut Paoli Calmette, Marseille
  - Montpellier - GCS Centre de Cancérologie du Grand Montpellier, Montpellier
  - CH de Mulhouse, Mulhouse
  - Nantes - ICO René Gauducheau, Nantes
  - Nevers - CH, Nevers
  - Centre Antoine Lacassagne, Nice
  - Orléans - Hôpital de la Source, Orléans
  - AP-HP Hopital Tenon - Pneumologie, Paris
  - Paris - APHP Bichat, Paris
  - Paris - APHP Saint-Louis, Paris
  - Pau - CH, Pau
  - Pontoise - CH, Pontoise
  - Centre Hospitalier, Saint-Quentin
  - Nouvel Hopital Civil - Pneumologie, Strasbourg
  - Centre Hospitalier Intercommunal, Toulon
  - HIA Saint Anne, Toulon
  - Tours - CHU, Tours
  - CH de Villefranche - Pneumologie, Villefranche
  - Villeneuve d'Ascq - Hôpital Privé, Villeneuve-d'Ascq

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Cortot AB, Madroszyk A, Giroux-Leprieur E, Molinier O, Quoix E, Berard H, Otto J, Rault I, Moro-Sibilot D, Raimbourg J, Amour E, Morin F, Hureaux J, Moreau L, Debieuvre D, Morel H, Renault A, Pichon E, Huret B, Charpentier S, Denis MG, Cadranel J. First-Line Afatinib plus Cetuximab for EGFR-Mutant Non-Small Cell Lung Cancer: Results from the Randomized Phase II IFCT-1503 ACE-Lung Study. Clin Cancer Res. 2021 Aug 1;27(15):4168-4176. doi: 10.1158/1078-0432.CCR-20-4604. Epub 2021 May 24. PMID 34031056
- See also: IFCT website — http://www.ifct.fr/index.php/fr/la-recherche/item/2032-ifct-1503-ace